CLINICAL TRIAL: NCT03827785
Title: The Efficacy and Safety of Repeated Transcranial Magnetic Stimulation for Treatment of Methamphetamine Dependence: a Multicenter, Double-blind, Randomized Controlled Clinical Trial
Brief Title: Transcranial Magnetic Stimulation for Treatment of Methamphetamine Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Wuxi Mental Health Center, Jiangsu Provence, China (Unknown); Suzhou Guangji Hospital, Jiangsu Provence, China (Unknown); Wuhan Mental Health Center, Hubei Provence, China (Unknown); Yunnan Institute For Drug Abuse (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HFJiang-002
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Methamphetamine-dependence
Keywords: repetitive transcranial magnetic stimulation (rTMS); randomized clinical trials; treatment; craving; cognitive function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS treatment group (Experimental): Stimulate the dorsal lateral prefrontal cortex with the iTBS pattern. The therapy will be conducted for 30 days.
  Interventions: Device: rTMS treatment group
- sham rTMS treatment group (Sham Comparator): Stimulate the dorsal lateral prefrontal cortex with the sham iTBS pattern and coil. The therapy will be conductedfor 30 days.
  Interventions: Device: sham rTMS treatment group

INTERVENTIONS:
Device: rTMS treatment group — For rTMS treatment, we will stimulate the dorsal lateral prefrontal cortex of each patients using the iTBS pattern everyday. Treatment will lasted for 30 days.
  Arms: rTMS treatment group
Device: sham rTMS treatment group — For sham rTMS treatment, we will stimulate the dorsal lateral prefrontal cortex of each patients using the sham iTBS pattern and sham coil everyday for 30 minutes. Treatment will lasted for 30 days.
  Arms: sham rTMS treatment group

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) was used to treat methamphetamine (MA) addiction in previous studies, while the evidence-based protocols still required. The aim of this research is to evaluating the effectiveness and safety of rTMS treatment in improving the days of abstinence maintenance. In addition, treatment effect on cognitive impairment, psychological craving and depression are also evaluated during the study.

DETAILED DESCRIPTION:
First, a multicenter, double-blind, randomized control study is going to be carried out. 100 recruited patients will be randomized assigned to the intervention group and the control group, receiving either 4-week of repetitive transcranial magnetic stimulation (rTMS) treatment or 4-week of sham rTMS treatment. Both groups will receive 12-week urine drug test follow-up (1 time per week). Negative rate of urine test during the follow-up period is set as primary outcome. Cognitive function, craving, depression are also evaluated before and after the intervention.

Secondly, another 40 patients will be recruited from these 100 patients (20 subjects each group). Magnetic resonance spectroscopy (MRS) test is applied to investigate the potential neurobiological mechanism of rTMS treatment. This study will be very helpful to develop an evidence-based rTMS treatment protocols for MA dependent patients and decrease risk of relapse for both the patients and their families.

ELIGIBILITY:
Inclusion Criteria:

1. In accordance with the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) for methamphetamine (MA) use disorders
2. Junior high school degree or above
3. Normal vision and hearing
4. Dextromanual
5. Less than one month before last drug use

Exclusion Criteria:

1. Have a disease that affect cognitive function such as history of head injury, cerebrovascular disease, epilepsy, etc
2. Have cognitive-promoting drugs in the last 6 months
3. Other substance abuse or dependence in recent five years (except nicotine)
4. Mental impairment, Intelligence Quotient (IQ) < 70
5. Mental disorders
6. Physical disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Negative rate urine test | 12 weeks
  After treatment, patients will be asked to participate urine test for 12 times once a week. Loss of visit or rejection for urine test will be treated as urine test positive.
  Negative rate of urine drug test = actual number of negative urine tests / 12.

SECONDARY OUTCOMES:
Change of Craving assessed by Visual Analog Scale | 12 weeks
  evaluate all participants' craving for for methamphetamine assessed by Visual Analog Scales (VAS). Score of VAS range from 0 to 10, and higher values represent high level of craving.
Cognitive function assessed by CogState Battery (CSB) | 12 weeks
  evaluate all participants' cognitive function by the computerized CogState Battery (CSB) Chinese version
Depression status assessed by Hamilton depression scale (HAMD-17) | 12 weeks
  Evaluate all participants' depression status by Hamilton depression scale (HAMD-17) HAMD can be summarized into 7 types of factor structure: (1) anxiety/somatization:; (2) weight: weight loss (3) Cognitive obstacles; (4) day and night changes; (5) Block; (6) sleep disorder; (7) feeling of despair. The total score can reflect the severity of the symptom, that is, The lighter the symptoms, the lower the score, and vice versa. Mild depression: HAMD 17 scores > 7 points, ≤ 17 points; moderate depression: HAMD 17 scores > 17 points, ≤ 24 points; severe depression: HAMD 17 scores > 24 points.

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Jiang, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Rehabilitation Center, Shanghai, China